CLINICAL TRIAL: NCT01379417
Title: Probiotics Supplementation and Nutritional Benefit in Premature Infants
Brief Title: Probiotics Supplementation in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 04.01.FR.INF; 2006-A00062-49 (Other: DIRECTION GENERALE DE LA SANTE)
Record Dates: First submitted 2011-05-10; First posted 2011-06-23 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Prematurity
Keywords: Prematurity; Nutrition; Growth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Maltodextrin (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Probiotic supplementation
- Probiotic B lactis/B longum (Active Comparator): Bifidobacterium lactis + Bifidobacterium longum
  Interventions: Dietary Supplement: Probiotic supplementation
- Probiotic B longum (Active Comparator): Bifidobacterium longum
  Interventions: Dietary Supplement: Probiotic supplementation
- Probiotic B lactis (Active Comparator): Bifidobacterium lactis
  Interventions: Dietary Supplement: Probiotic supplementation

INTERVENTIONS:
Dietary Supplement: Probiotic supplementation — 1 capsule per day, from inclusion to 4 or 6 weeks after inclusion

SUMMARY:
The main objective is to assess the nutritional benefit of probiotics supplementation on premature infants growth. As secondary objectives, different parameters related to probiotics tolerance will be measured.

ELIGIBILITY:
Inclusion criteria

* Gestational age between 26 weeks and 31 weeks
* Birth weight between 700 to 1600 g
* Eutrophic infants (weight between -2 to 2 DS, Usher curves)
* Admitted to one of the participating hospital unit within the 8 days following the birth, the birth date equals the 1st day of life.
* Still on parenteral feeding or infusion on the 5th day of birth

Non inclusion criteria

* Digestive disorders > or equal to 1b on Bell stage
* Severe intra-ventricular haemorrhage (stage 3-4) before 5th day of life.
* Severe malformations or digestive malformations
* No antenatal corticosteroid therapy
* Severe medical or surgical disorder affecting the absorption, digesting and as a result the growth (Hirschsprung disease, lactose intolerance, cow milk protein allergy, mucoviscidosis).
* Parents geographical distance preventing the hospitalization follow-up in the hospital participating unit (geographical distance planned before the infant reaches 1500 g or 32 weeks of gestational age)

Exclusion criteria

* Enteral/Oral feeding termination during more than 72 hours due to severe digestive disorders (> or equal to 2a on Bell stage )
* Serious digestive surgery

Ages: 1 Day to 8 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 199 (Actual)
Dates: Start 2007-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Weight (g) | From 4 to 6 weeks after inclusion

SECONDARY OUTCOMES:
Growth | between inclusion date and 4 to 6 weeks after inclusion (= end of supplementation period)
  measured by:
  * weight gain (g/day)
  * height (cm/week)
  * head circumference(cm/week)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Picaud, Pr, Principal Investigator — Hôpital de la Croix-Rousse
Locations (3):
- France (3):
  - Service de Nénatologie, Hôpital Femme Mère Enfant, Bron
  - Service de Réanimation Néonatale et Néonatologie, Hôpital de la Croix Rousse, Lyon
  - Service de Réanimation Néonatale, Hôpital Arnaud de Villeneuve, Montpellier

REFERENCES:
- [Derived] Hays S, Jacquot A, Gauthier H, Kempf C, Beissel A, Pidoux O, Jumas-Bilak E, Decullier E, Lachambre E, Beck L, Cambonie G, Putet G, Claris O, Picaud JC. Probiotics and growth in preterm infants: A randomized controlled trial, PREMAPRO study. Clin Nutr. 2016 Aug;35(4):802-11. doi: 10.1016/j.clnu.2015.06.006. Epub 2015 Jul 16. PMID 26220763